CLINICAL TRIAL: NCT00929331
Title: Immunogenicity and Safety Study of GSK Biologicals' Trivalent Split Virion Influenza Vaccine Fluviral® (2009 - 2010 Season) in Adults Aged 18 to 60 Years and Over 60 Years.
Brief Title: Immunogenicity & Safety Study of Fluviral® (2009 - 2010 Season) in Adults Aged 18 to 60 Years and Over 60 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 110586
Record Dates: First submitted 2009-06-25; First posted 2009-06-29 (Estimated); Results first posted 2010-08-13 (Estimated); Last update posted 2020-11-09 (Actual); Status verified 2020-10

CONDITIONS: Influenza, Human
Keywords: Influenza; Fluviral®
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

ARMS (2):
- Fluviral Adult Group (Experimental): Subjects aged between 18 and 60 years who received one dose of Fluviral® (2009-2010 season) intramuscularly in the deltoid region of the non-dominant arm
  Interventions: Biological: Fluviral®
- Fluviral Elderly Group (Experimental): Subjects over 60 years of age who received one dose of Fluviral ® (2009-2010 season) intramuscularly in the deltoid region of the non-dominant arm
  Interventions: Biological: Fluviral®

INTERVENTIONS:
Biological: Fluviral® — Intramuscular injection, one dose

SUMMARY:
This study is designed to test the safety and immunogenicity of Fluviral® (2009 - 2010 Season) in adults aged 18 to 60 years and over 60 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject
* Male and female adults, 18 to 60 years of age and over 60 years of age.
* Satisfactory baseline medical assessment by history and physical examination
* Comprehension of the study requirements, ability to comprehend and comply with procedures for collection of safety data, expressed availability for the required study period, and ability and willingness to attend scheduled visits.
* Female subjects of non-childbearing potential may be enrolled in the study.

  * Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Participation in previous year's (2008) Fluviral® registration study
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s)/product(s) within 30 days preceding the first dose of study vaccine/product, or planned use during the study period.
* Acute disease at the time of enrollment. All vaccines can be administered to persons with a minor illness such as diarrhea, mild upper respiratory infection with or without low-grade febrile illness, i.e. oral temperature <38.0°C.
* Significant acute or chronic, uncontrolled medical or psychiatric illness. "Uncontrolled" is defined as:

Requiring institution of new medical or surgical treatment within one (1) month prior to study enrollment, or Requiring the re-institution of a previously discontinued medication or medical treatment within one month prior to study enrollment, or Requiring a change in medication dosage in the one month prior to study enrollment due to uncontrolled symptoms or drug toxicity (elective dosage adjustments in stable subjects are acceptable), or Hospitalization or an event fulfilling the definition of a SAE within one month prior to study enrollment.

• Any confirmed or suspected immunosuppressive condition including: History of human immunodeficiency virus (HIV) infection, Cancer or treatment for cancer, within 3 years of study enrollment. Persons with a history of cancer who are disease-free without treatment for 3 years or more are eligible.

* History of renal impairment.
* History of hepatic dysfunction due to hepatitis B, C or toxins including alcohol.
* Complicated insulin-dependent diabetes mellitus.
* Unstable cardiopulmonary disease requiring chronic medical therapy or associated with functional impairment.
* Presence of blood dyscrasias, including hemoglobinopathies and myelo- or lymphoproliferative disorder.
* Receipt of systemic glucocorticoids within 1 month of study enrollment, or any cytotoxic or immunosuppressive drugs within six months of study enrollment. Inhaled and topical steroids are allowed.
* A history of any demyelinating disease including Multiple Sclerosis and Guillain-Barré syndrome.
* Presence of an active neurological disorder.
* History of chronic alcohol consumption and/or drug abuse.
* Any significant disorder of coagulation that increases the risk of intramuscular injections or treatment with coumadin derivatives or heparin. Persons receiving prophylactic antiplatelet medications, e.g. low-dose aspirin, and without a clinically-apparent bleeding tendency are eligible.
* Receipt of an influenza vaccine within 6 months prior to study enrollment.
* Administration of any vaccines within 30 days prior to study enrollment or during the study period. Subjects who receive such treatment after enrollment will be followed per protocol and included in the safety analysis, but excluded from the according-to-protocol cohort.
* Administration of immunoglobulins and/or any blood products within the three months preceding the administration of the study vaccine or planned during the study.
* Any known or suspected allergy to any constituent of Fluviral® and/or a history of anaphylactic type reaction to constituent of the vaccine.
* A history of severe adverse reaction to a previous influenza vaccination.
* Lactating/nursing female.
* Any condition which, in the opinion of the investigator, prevents the subject from participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2009-07-11 (Actual); Primary Completion 2009-08-01 (Actual); Study Completion 2009-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 110586 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110586 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 110586 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110586 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 110586 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 110586 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110586 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fluviral Adult Group | Fluviral Elderly Group
Started | 55 | 55
Completed | 55 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluviral Adult Group | Fluviral Elderly Group | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.1 (14.83) | 66.8 (4.10) | 51.0 (19.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 31 | 63
  Male | 23 | 24 | 47

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of Hemagglutination Inhibition (HI) Antibodies
Description: Data are displayed as GMTs for each of the three influenza virus vaccine strains: A/Brisbane(H1N1); A/Uruguay(H3N2); B/Brisbane.
Time Frame: At Day 0
Population: Analysis was performed on the According-To-Protocol (ATP) Cohort for immunogenicity which included all evaluable subjects for whom data concerning immunogenicity outcome variables were available. These included subjects for whom assay results were available for antibodies against at least on study vaccine antigen component after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Fluviral Adult Group | Fluviral Elderly Group
Number analyzed (Participants) | 55 | 55
titer
  A/Brisbane | 27.2 [18.8 to 39.5] | 22.8 [16.8 to 31.1]
  A/Uruguay | 33.3 [21.8 to 50.7] | 45.9 [31.3 to 67.3]
  B/Brisbane | 36.8 [26.5 to 51.1] | 48.3 [34.4 to 67.7]

2. Primary Outcome: GMTs of HI Antibodies
Description: as for outcome 1
Time Frame: At Day 21 after vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Fluviral Adult Group | Fluviral Elderly Group
Number analyzed (Participants) | 55 | 55
titer
  A/Brisbane | 139.2 [101.6 to 190.6] | 40.2 [29.7 to 54.5]
  A/Uruguay | 273.3 [192.8 to 387.3] | 141.0 [100.0 to 198.8]
  B/Brisbane | 230.6 [177.4 to 299.7] | 131.5 [95.2 to 181.7]

3. Primary Outcome: Number of Subjects With a Serum HI Titer Equal to or Above the Cut-off Value
Description: The cut-off value was defined as a serum HI titer >= 1:40, which is usually accepted as indicating protection. Data are displayed for each of the three influenza virus vaccine strains: A/Brisbane(H1N1); A/Uruguay(H3N2); B/Brisbane.
Time Frame: At Day 0
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Fluviral Adult Group | Fluviral Elderly Group
Number analyzed (Participants) | 55 | 55
subjects
  A/Brisbane | 27 | 18
  A/Uruguay | 23 | 32
  B/Brisbane | 31 | 38

4. Primary Outcome: Number of Subjects With a Serum HI Titer Equal to or Above the Cut-off Value
Description: as for outcome 3
Time Frame: At Day 21 after vaccination
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Fluviral Adult Group | Fluviral Elderly Group
Number analyzed (Participants) | 55 | 55
subjects
  A/Brisbane | 51 | 27
  A/Uruguay | 54 | 50
  B/Brisbane | 55 | 51

5. Primary Outcome: Number of Seroconverted Subjects
Description: A seroconverted subject is a subject who had either a prevaccination titer < 1:10 and a post-vaccination titer >= 1:40 or a pre-vaccination titer >= 1:10 and at least a four-fold increase in post-vaccination titer. Data are displayed for each of the three influenza virus vaccine strains: A/Brisbane(H1N1); A/Uruguay(H3N2); B/Brisbane.
Time Frame: At Day 21 after vaccination
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Fluviral Adult Group | Fluviral Elderly Group
Number analyzed (Participants) | 55 | 55
subjects
  A/Brisbane | 26 | 8
  U/Uruguay | 35 | 17
  B/Brisbane | 38 | 17

6. Primary Outcome: Seroconversion Factors
Description: Seroconversion factors are defined as the fold increase in serum HI GMTs post-vaccination (Day 21) compared to pre-vaccination (Day 0). Data are displayed for each of the three influenza virus vaccine strains: A/Brisbane(H1N1); A/Uruguay(H3N2); B/Brisbane.
Time Frame: At Day 21 after vaccination
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Fluviral Adult Group | Fluviral Elderly Group
Number analyzed (Participants) | 55 | 55
ratio
  A/Brisbane | 5.1 [3.3 to 8.0] | 1.8 [1.4 to 2.2]
  U/Uruguay | 8.2 [5.4 to 12.5] | 3.1 [2.2 to 4.3]
  B/Brisbane | 6.3 [4.5 to 8.8] | 2.7 [2.0 to 3.7]

7. Primary Outcome: Number of Subjects With a Pre-vaccination Titer Below the Cut-off Value and a Post-vaccination Titer Equal to or Above the Cut-off Value
Description: The cut-off value was a titer of 1:40. Data are displayed for each of the three influenza virus vaccine strains: A/Brisbane(H1N1); A/Uruguay(H3N2); B/Brisbane.
Time Frame: At Day 21 after vaccination
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Fluviral Adult Group | Fluviral Elderly Group
Number analyzed (Participants) | 32 | 37
subjects
  A/Brisbane: number analyzed (Participants) | 28 | 37
  A/Brisbane | 24 | 9
  A/Uruguay: number analyzed (Participants) | 32 | 23
  A/Uruguay | 31 | 18
  B/Brisbane: number analyzed (Participants) | 24 | 17
  B/Brisbane | 24 | 13

8. Secondary Outcome: Number of Subjects Reporting Any Solicited Local Symptoms
Description: Solicited local symptoms assessed include pain, redness and swelling at the site of injection. Any = Solicited local symptoms are presented regardless of their intensity grade
Time Frame: During a 4-day (Day 0-3) follow-up period after vaccination
Population: Analysis was performed on the Total Vaccinated Cohort, which included all subjects for whom data were available.
Measure: Number; unit: subjects
Arm/Group | Fluviral Adult Group | Fluviral Elderly Group
Number analyzed (Participants) | 55 | 55
subjects
  Pain | 34 | 16
  Redness | 1 | 0
  Swelling | 2 | 1

9. Secondary Outcome: Number of Subjects Reporting Grade 3 Solicited Local Symptoms
Description: Solicited local symptoms assessed include pain, redness and swelling at the site of injection. Grade 3 pain = pain that prevented normal activity, Grade 3 redness/swelling = redness/swelling > 100 mm
Time Frame: During a 4-day (Day 0-3) follow-up period after vaccination
Population: Analysis was performed on the Total Vaccinated Cohort, which included all subjects for whom data were available.
Measure: Number; unit: subjects
Arm/Group | Fluviral Adult Group | Fluviral Elderly Group
Number analyzed (Participants) | 55 | 55
subjects
  Pain | 1 | 0
  Redness | 0 | 0
  Swelling | 0 | 0

10. Secondary Outcome: Number of Subjects Reporting Any Solicited General Symptoms
Description: Solicited local symptoms assessed include bronchospasm, chills, cough, fatigue, headache, joint pain at other location, muscle aches, red eyes, sore throat, swelling of the face, temperature (orally) in degrees celsius. Any = solicited general symptoms are presented regardless of their intensity grade or relationship to vaccination. For temperature this means equal to or above 38.0 degrees celsius.
Time Frame: During a 4-day (Day 0-3) follow-up period after vaccination
Population: Analysis was performed on the Total Vaccinated Cohort, which included all subjects for whom data were available.
Measure: Number; unit: subjects
Arm/Group | Fluviral Adult Group | Fluviral Elderly Group
Number analyzed (Participants) | 55 | 55
subjects
  Bronchospasm | 2 | 0
  Chills | 5 | 5
  Cough | 4 | 3
  Fatigue | 11 | 7
  Headache | 7 | 6
  Joint pain at other location | 5 | 3
  Muscle aches | 10 | 8
  Red eyes | 1 | 0
  Sore throat | 2 | 2
  Swelling of the face | 0 | 0
  Temperature | 1 | 0

11. Secondary Outcome: Number of Subjects Reporting Grade 3 Solicited General Symptoms
Description: Solicited local symptoms assessed include bronchospasm, chills, cough, fatigue, headache, joint pain at other location, muscle aches, red eyes, sore throat, swelling of the face, temperature (orally) in degrees celsius. Grade 3 general symptom = symptom that prevented normal activity Grade 3 temperature = temperature above 39.0 degrees celsius
Time Frame: During a 4-day (Day 0-3) follow-up period after vaccination
Population: Analysis was performed on the Total Vaccinated Cohort, which included all subjects for whom data were available.
Measure: Number; unit: subjects
Arm/Group | Fluviral Adult Group | Fluviral Elderly Group
Number analyzed (Participants) | 55 | 55
subjects
  Bronchospasm | 0 | 0
  Chills | 0 | 0
  Cough | 0 | 0
  Fatigue | 0 | 1
  Headache | 0 | 0
  Joint pain at other location | 0 | 0
  Muscle aches | 0 | 0
  Red eyes | 0 | 0
  Sore throat | 0 | 0
  Swelling of the face | 0 | 0
  Temperature | 0 | 0

12. Secondary Outcome: Number of Subjects Reporting Related Solicited General Symptoms
Description: Solicited local symptoms assessed include bronchospasm, chills, cough, fatigue, headache, joint pain at other location, muscle aches, red eyes, sore throat, swelling of the face, temperature (orally) in degrees celsius. Related = general symptom assessed by the investigator as related to the vaccine
Time Frame: During a 4-day (Day 0-3) follow-up period after vaccination
Population: Analysis was performed on the Total Vaccinated Cohort, which included all subjects for whom data were available.
Measure: Number; unit: subjects
Arm/Group | Fluviral Adult Group | Fluviral Elderly Group
Number analyzed (Participants) | 55 | 55
subjects
  Bronchospasm | 2 | 0
  Chills | 5 | 5
  Cough | 4 | 3
  Fatigue | 11 | 7
  Headache | 7 | 6
  Joint pain at other location | 5 | 3
  Muscle aches | 10 | 8
  Red eyes | 1 | 0
  Sore throat | 2 | 2
  Swelling of the face | 0 | 0
  Temperature | 1 | 0

13. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs)
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any = unsolicited adverse event regardless of intensity. Grade 3 = unsolicited AE that prevented normal activity Related = unsolicited AE assessed by the investigator as related to the vaccination.
Time Frame: During a 21-day (Day 0-20) follow-up period after vaccination
Population: Analysis was performed on the Total Vaccinated Cohort, which included all subjects for whom data were available.
Measure: Number; unit: subjects
Arm/Group | Fluviral Adult Group | Fluviral Elderly Group
Number analyzed (Participants) | 55 | 55
subjects
  Any | 13 | 4
  Grade 3 | 1 | 0
  Related | 3 | 0

14. Secondary Outcome: Number of Subjects With Serious Adverse Events
Description: SAEs assessed include medical occurrences that result in death, is life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: From the beginning up to the end of the study (Day 0 - Day 21)
Measure: Number; unit: subjects
Arm/Group | Fluviral Adult Group | Fluviral Elderly Group
Number analyzed (Participants) | 55 | 55
subjects | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited adverse events were collected during the 4-day (Day 0-3) post-vaccination period, unsolicited and serious adverse events were collected during the 21-day (Day 0-20) post-vaccination period.
Description: For this study, the Total Number (#) of Participants Affected by Other (non-serious) Adverse Events (AEs) was analyzed separately for expected AEs and for unexpected AEs. A consolidated analysis of all expected and unexpected AEs was not technically possible to be performed and the relevant data are no longer available. Therefore, the Total #Participants Affected in Other Adverse Events Table is currently populated by the highest value of #Participants affected within other AE's table.
Arm/Group | Fluviral Adult Group | Fluviral Elderly Group
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55
Other Adverse Events (participants affected / at risk) | 34/55 | 16/55
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fluviral Adult Group (N=55) | Fluviral Elderly Group (N=55)
Pain (General disorders) | 34 | 16
chills (General disorders) | 5 | 5
Cough (General disorders) | 4 | 3
Fatigue (General disorders) | 11 | 7
Headache (General disorders) | 7 | 6
Joint pain at other location (General disorders) | 5 | 3
Muscle aches (General disorders) | 10 | 8
Headache (Nervous system disorders) | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.